CLINICAL TRIAL: NCT07097324
Title: Effectiveness of an Interactive Video- and Game-Based Oral Health Education Intervention Among 11-Year-Old Schoolchildren in Pulau Pinang: A Cluster Randomised Controlled Trial
Brief Title: Interactive Video- and Game-Based Oral Health Education for 11-Year-Old Schoolchildren
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Stephanie Oung Ker Yue, Doctoral Candidate, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: USM/JEPeM/KK/25030264; NMRR ID-25-01175-JV3 (Registry Identifier: National Medical Research Register)
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Oral Health
Keywords: Education, Dental; Health Knowledge, Attitudes, Practice; Oral Hygiene; Oral Health; Child
MeSH Terms: conditions — Behavior | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video- and Game-Based Oral Health Education (Experimental): Participants in the intervention group will receive three video- and game-based oral health education sessions, each delivered one week apart by the principal investigator, in addition to the conventional oral health talk provided through the school dental service.
  Interventions: Behavioral: Video- and Game-Based Oral Health Education; Behavioral: Conventional Oral Health Talk
- Conventional Oral Health Talk (Active Comparator): Participants in the control group will receive a conventional oral health talk provided through the school dental service.
  Interventions: Behavioral: Conventional Oral Health Talk

INTERVENTIONS:
Behavioral: Video- and Game-Based Oral Health Education — A video- and game-based oral health education intervention will be delivered to the participants in the intervention group over three weekly sessions. In the first session, participants will watch a video that highlights key messages on oral health, including the importance of oral health, the consequences of poor oral health and recommended oral health practices. This will be followed by an interactive quiz to reinforce the content of the video. In the second session, a video demonstrating proper tooth brushing and flossing techniques will be shown. Participants will then practice these techniques using tooth models. The third session will feature a video on cariogenic food consumption, followed by an interactive educational game in which participants identify non-cariogenic foods.
  Arms: Video- and Game-Based Oral Health Education
Behavioral: Conventional Oral Health Talk — A conventional oral health talk will be delivered to participants in both the control and intervention groups. The talk will cover key messages on oral health, including the importance of oral health, consequences of poor oral health and recommended oral health practices.

SUMMARY:
The goal of this cluster randomised controlled trial is to learn if an interactive video- and game-based oral health education intervention helps improve oral health outcomes among 11-year-old schoolchildren in Pulau Pinang, Malaysia. The main questions it aims to answer are:

* Does the intervention improve oral hygiene status?
* Does the intervention improve oral health knowledge, attitudes and hygiene practices?
* Does the intervention reduce the frequency of consuming foods that can cause tooth decay (cariogenic foods)?

Investigators will compare a group that receives the video- and game-based oral health education intervention along with a conventional oral health talk to a group that receives only the conventional oral health talk. This will help determine whether the video- and game-based oral health education intervention is more effective than the conventional oral health talk alone.

Participants will:

* Receive either three weekly sessions of the video- and game-based oral health education intervention in addition to a conventional oral health talk, or only the conventional oral health talk.
* Take part in assessments, including a clinical examination to check oral hygiene status and a self-administered questionnaire on oral health knowledge, attitudes, hygiene practices and frequency of cariogenic food consumption. These assessments will take place at three time points: before the intervention, one month after and three months after the intervention is completed.

DETAILED DESCRIPTION:
This is a two-arm, parallel-group, single-blinded, cluster randomised controlled trial evaluating the effectiveness of an interactive video- and game-based oral health education intervention among 11-year-old schoolchildren in Pulau Pinang, Malaysia.

The allocation follows a 1:1 ratio. One district will be randomly selected and assigned to the intervention group, and another to the control group, using computer-generated random numbers in IBM SPSS Statistics for Windows, Version 29. Within each district, two government national primary schools will be randomly selected, and from each school, two classes will be randomly chosen. All eligible students in the selected classes, with written parental/guardian consent and written participant assent, will be included.

The control group will receive a conventional oral health talk provided through the school dental service. The intervention group will receive three weekly video- and game-based oral health education sessions delivered by the principal investigator, in addition to the conventional oral health talk.

Assessments will be conducted at three time points: pre-intervention, one month post-intervention and three months post-intervention. The primary outcome is oral hygiene status, while secondary outcomes include oral health knowledge, oral health attitudes, oral hygiene practices and frequency of cariogenic food consumption. Oral hygiene status will be assessed by a calibrated clinician using the Simplified Debris Index (DI-S) while secondary outcomes will be assessed using a validated self-administered questionnaire. The trial is single-blinded, with clinical examiners blinded to group allocation.

Sample size was calculated using G*Power software version 3.1.9.7 for repeated measures Analysis of Variance (ANOVA) (between factors). Assuming an effect size of 0.25, α = 0.05, power = 0.8 and a correlation of 0.5 among repeated measures, the required sample size is 86 participants. After adjusting for a 20% attrition rate and a design effect of 2 for cluster randomisation, the final sample size is 216 participants (108 per group).

All data will be analysed using IBM SPSS Statistics for Windows, Version 29. Descriptive statistics will summarise the data. Pre-intervention between-group comparisons will be conducted using the Pearson chi-square tests for categorical variables and independent t-tests for numerical variables. Mixed ANOVA will be used to assess and compare oral hygiene status, oral health knowledge, oral health attitudes, oral hygiene practices and frequency of cariogenic food consumption within and between the intervention and control groups at various time points (pre-intervention, one month post-intervention and three months post-intervention). If needed, mixed Analysis of Covariance (ANCOVA) will be performed to adjust for potential confounding factors. When significant effects are observed, post-hoc pairwise comparisons will be conducted to identify specific time points with significant differences. A significance level of p<0.05 will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Schoolchildren who are Malaysian citizens.
* Schoolchildren born in year 2014.
* Schoolchildren studying at government national primary schools under the Ministry of Education Malaysia.
* Schoolchildren who are able to understand, read and write in Malay language.

Exclusion Criteria:

* Schoolchildren with underlying chronic medical conditions.
* Schoolchildren wearing intra-oral appliances.
* Schoolchildren with learning or intellectual disabilities.
* Schoolchildren with impaired manual dexterity.
* Schoolchildren with visual or hearing impairments.

Ages: 11 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2025-08-04 (Actual); Primary Completion 2025-12-05 (Actual); Study Completion 2025-12-05 (Actual)

PRIMARY OUTCOMES:
Change in Oral Hygiene Status Assessed Using the Simplified Debris Index (DI-S) | Pre-Intervention, One Month Post-Intervention and Three Months Post-Intervention
  The Simplified Debris Index (DI-S), a component of the Simplified Oral Hygiene Index, will be used to assess the change in oral hygiene status. Six tooth surfaces-buccal of upper and lingual of lower first molars, and labial of upper right and lower left central incisors-will be examined. A no. 5 dental explorer will be used to detect debris, scored as follows: 0 = No debris or stain present; 1 = Soft debris covering not more than one third of the tooth surface being examined or the presence of extrinsic stains without debris regardless of surface area covered; 2 = Soft debris covering more than one third but not more than two thirds of the exposed tooth surface; 3 = Soft debris covering more than two thirds of the exposed tooth surface. The debris scores will be totaled and divided by the number of surfaces assessed to obtain the average score (DI-S), which is classified as 'good' (0-0.6), 'fair' (0.7-1.8) or 'poor' (1.9-3.0).

SECONDARY OUTCOMES:
Change in Oral Health Knowledge, Attitudes and Hygiene Practices Assessed Using a Self-Administered Questionnaire Adapted from the Health Promotion Questionnaire Index (HPQI) | Pre-Intervention, One Month Post-Intervention and Three Months Post-Intervention
  Oral health knowledge, attitudes and hygiene practices will be assessed using a validated self-administered questionnaire adapted from the Health Promotion Questionnaire Index (HPQI). The knowledge domain has 11 positively worded items rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree), with total scores ranging from 11 to 55. The attitude domain includes 15 items rated on a 4-point Likert scale (1 = strongly disagree to 4 = strongly agree). Items 1 to 12 are positively worded, while items 13 to 15 are negatively worded and reverse scored. Total scores range from 15 to 60. The hygiene practice domain has 4 items with 'Yes' or 'No' responses, scored as 1 and 0, respectively. Total scores range from 0 to 4. Scores for knowledge, attitude and hygiene practice will be converted into percentages and categorised as 'poor' (<60%), 'moderate' (60%-79%) or 'good' (80%-100%).
Change in Frequency of Cariogenic Food Consumption Assessed Using the Self-Administered Malay-Language Cariogenic Food Frequency Questionnaire (M-CFFQ) | Pre-Intervention, One Month Post-Intervention and Three Months Post-Intervention
  Frequency of cariogenic food consumption will be assessed using the self-administered Malay-Language Cariogenic Food Frequency Questionnaire (M-CFFQ). Originally developed for parental reporting, the M-CFFQ has been validated for self-administration by 11-year-old schoolchildren. It includes 37 food items across 15 different types of cariogenic foods. Responses range from 'never/rarely' to '2 to 3 times daily', scored from 1 to 7. The total cariogenic food frequency (CFF) score, ranging from 37 to 259, is calculated by summing the scores of all items; higher scores indicate more frequent consumption of cariogenic food. CFF scores for individual food items are also calculated using a weighted formula based on response percentages and scale ratings. Food items are then categorised as 'least consumed' (0%-29.9%), 'moderately consumed' (30.0%-79.9%), or 'highly consumed' (80.0%-100%).

CONTACTS AND LOCATIONS:
Locations (1):
- Pulau Pinang State Education Department, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No
Data can be shared upon reasonable request and in accordance with applicable data protection regulations.